CLINICAL TRIAL: NCT02844231
Title: Functional Imagery of Sleepwalking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UF 8585
Record Dates: First submitted 2016-07-18; First posted 2016-07-26 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Sleepwalking
MeSH Terms: conditions — Somnambulism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sleepwalker, SW episode (Other): Sleepwalker patients undergo single-photon emission computed tomography during a sleepwalking episode.
  Interventions: Other: Single-photon emission computed tomography
- Sleepwalkers, slow wave sleep (Other): Sleepwalker patients undergo single-photon emission computed tomography during slow-wave sleep.
  Interventions: Other: Single-photon emission computed tomography
- Control group (Other): Control subjects undergo single-photon emission computed tomography during slow-wave sleep.
  Interventions: Other: Single-photon emission computed tomography

INTERVENTIONS:
Other: Single-photon emission computed tomography

SUMMARY:
Sleepwalking (also called somnambulism) is a disorder in which only SWS is disrupted. This NREM parasomnia is characterized by inappropriate motor behaviors, usually initiated during arousal from SWS, that induce psychological distress and alter quality of life, leading to fatigue, excessive daytime sleepiness, and objectively impaired vigilance in the morning.

The pathophysiology of sleepwalking remains poorly understood. Sleepwalkers had difficulty maintaining stable, consolidated sleep and experienced more arousals and microarousals, specifically from SWS, leading to increased NREM instability, especially during the first sleep cycles. The brain is partially awake, resulting in behavioral manifestations, and partially in NREM sleep, resulting in no conscious awareness of actions.

A Single Photonic Emission Computed Tomography (SPECT) study of one sleepwalking episode found increased activation in the posterior cingulate cortex and cerebellum, with deactivation in the frontoparietal associative cortices. Data from intracerebral EEGs during confusional arousals confirmed both local arousal of the motor and cingulate cortices and increased delta activity in the frontoparietal associative cortices.

The investigators thus proposed a controlled study of SPECT imagery in 24 sleepwalkers (12 SPECT during a SW episode and 12 SPECT during slow wave sleep and 24 during wakefulness) and 12 controls (during slow wave sleep and wakefulness). SW episodes will be elicited by sleep deprivation condition associated with forced arousal (auditory stimulus).

The comparative analyses of SPECT acquisitions between different states (wakefulness, slow wave sleep and SW) and populations (sleepwalkers versus controls) will provide new insights about the complex pathophysiology of SW episodes.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Subject diagnosed with NREM parasomnia according the international classification of sleep disorders
* More than one episode per week
* More than one hypersynchronous delta wave arousal recorded on polysomnographic assessment
* Affiliated to social security
* Age between 18 years-old and 39 years-old

Exclusion Criteria:

* Patient taking any psychotropic drug during the two weeks before the inclusion
* Patient with obstructive sleep apnea Syndrome, restless legs syndrome, nocturnal epilepsy and unstable psychiatric disease.

CONTROL GROUP

Inclusion Criteria:

* Affiliated to social security
* Age between 18 years-old and 39 years-old

Exclusion Criteria:

* Subject taking psychotropic drug during the two weeks before the inclusion
* Subject with following medical history : NREM parasomnia, neurologic or psychiatric disorder, obstructive sleep apnea syndrome, restless legs syndrome, nocturnal epilepsy.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Brain metabolism measurement with brain scintigraphy | Day 0

SECONDARY OUTCOMES:
Cortical excitability measurement with transcranial magnetic stimulation | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France